CLINICAL TRIAL: NCT00461539
Title: Reducing Health Risk Behavior and Improving Health in Adolescent Depression
Brief Title: Reducing Health Risk Behavior and Improving Health in Adolescents With Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kaiser Permanente Research Foundation (Unknown)
Responsible Party: Principal Investigator, Joan Asarnow, Professor of Psychiatry & Biobehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH078596 (NIH); R01MH078596 (NIH); DAHBR 96-BHB
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2013-06

CONDITIONS: Depression; Adolescent Health
Keywords: Tobacco Use; Alcohol and Drug Use; Obesity; Risky Sexual Behavior
MeSH Terms: conditions — Depression; Tobacco Use; Obesity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Participants will receive treatment as usual
  Interventions: Other: Treatment as usual
- 1 (Experimental): Participants will receive the behavioral health intervention
  Interventions: Behavioral: Behavioral health intervention

INTERVENTIONS:
Other: Treatment as usual — Those participants receiving standard care will be referred to special programs as needed to reduce their involvement in risky health behaviors.
  Arms: 2
Behavioral: Behavioral health intervention — Participants assigned to the health education intervention will attend 10 weekly education sessions that will be led by trained health educators. Parents or guardians may be asked to attend sessions depending on their interest in the intervention and the age of the youth participant. Topics covered will include teenage smoking, alcohol and drug abuse, risky sexual behaviors, and obesity. Cognitive-behavioral strategies, role playing, and media clips will be used to stimulate discussion and involvement in the intervention.
  Arms: 1

SUMMARY:
This study will determine the effectiveness of a health education intervention in reducing health risk behavior and improving health in adolescents with depression.

DETAILED DESCRIPTION:
Depression is a common disorder among adolescents. If left untreated, it can cause significant disability, illness, and even death. Teens with depression often engage in risky health behaviors, such as smoking, drug and alcohol use, unprotected sex, and unhealthy eating and exercise patterns. By reducing these health risk behaviors, depressed adolescents may be able to avoid negative health consequences and improve their physical and mental health. This study will determine the effectiveness of a health education intervention in reducing risky health behaviors in adolescents with depression.

Participants in this study will be invited to enroll during a visit to a participating primary care clinic. Participants will be randomly assigned to either partake in a health education intervention or receive standard care. Both groups will continue to receive treatment through their primary care clinic. Those participants receiving standard care will be referred to special programs as needed to reduce their involvement in risky health behaviors. Participants assigned to the health education intervention will attend 10 weekly education sessions that will be led by trained health educators. Parents or guardians may be asked to attend sessions depending on their interest in the intervention and the age of the youth participant. Topics covered will include teenage smoking, alcohol and drug abuse, risky sexual behaviors, and obesity. Cognitive-behavioral strategies, role playing, and media clips will be used to stimulate discussion and involvement in the intervention. The intervention will be tailored to target the specific risky behaviors in which each participant engages. Motivational interviewing will also be used to build positive attitudes to support behavior change. All participants will attend follow-up visits to assess behavior change at Months 6 and 12 following study entry.

ELIGIBILITY:
Inclusion Criteria:

* CIDI diagnosis of major depression or probable depression based on youth self report
* Availability of a family member to provide informed consent

Exclusion Criteria:

* Lacks contact information (e.g., address, telephone number)
* Any functioning deficits or other characteristics that might interfere with study participation
* Currently in a living situation that might interfere with study participation (e.g., lives over 1 hour away from the study site)
* Lacks family available to participate in the intervention
* Mental retardation
* Does not speak English or Spanish

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 217 (Actual)
Dates: Start 2007-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Composite health risk behavior score | Measured at Months 6 and 12

SECONDARY OUTCOMES:
Composite International Diagnostic Interview (CIDI) depression diagnosis | Measured at Months 6 and 12
Satisfaction with care, as measured by the SF-12 health survey | Measured at Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Joan Asarnow, PhD, Principal Investigator — University of California, Los Angeles, Semel Institute of Neuroscience and Human Behavior
Locations (2):
- United States (2):
  - University of California, Los Angeles, Semel Institute for Neuroscience and Human Behavior, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California

REFERENCES:
- [Background] Bai S, Zeledon LR, D'Amico EJ, Shoptaw S, Avina C, LaBorde AP, Anderson M, Fitzpatrick OM, Asarnow JR. Reducing Health Risk Behaviors and Improving Depression in Adolescents: A Randomized Controlled Trial in Primary Care Clinics. J Pediatr Psychol. 2018 Oct 1;43(9):1004-1016. doi: 10.1093/jpepsy/jsy048. PMID 30016473
- [Background] Asarnow JR, Zeledon LR, D'Amico E, LaBorde A, Anderson M, Avina C, Arslanian T, Do MC, Harwood J, Shoptaw S. Depression and Health Risk Behaviors: Towards Optimizing Primary Care Service Strategies for Addressing Risk. Prim Health Care. 2014 Mar 1;4(1):152. doi: 10.4172/2167-1079.1000152. PMID 25309826